CLINICAL TRIAL: NCT01539421
Title: The Use of Home Exercise Program Based on Interactive Entertainment Computer System in Patients With Moderate to Severe COPD: Its Feasibility and Effects on Exercise Performance, Physical Activity, Dyspnea, and Quality of Life
Brief Title: Use of Wii Home Computer in Patients With Chronic Obstructive Pulmonary Disease: Effects on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trinity Health Of New England (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-06-007
Record Dates: First submitted 2012-02-21; First posted 2012-02-27 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: COPD
Keywords: COPD; exercise endurance
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exercise Intervention (Experimental): Use of Wii computer for enhanced exercise in COPD patients.
  Interventions: Behavioral: Use of Home exercise computer program

INTERVENTIONS:
Behavioral: Use of Home exercise computer program — After a 30-minute rest period the study patient performed a series of 4 representative exercises from the Wii under direct supervision by an investigator. Five minutes' rest was allotted between each exercise. The patient was instructed to exercise at his/her own pace, with a maximal duration of 5 minutes per exercise. The Oxycon Mobile was worn throughout this exercise, and the metabolic measurements listed above were recorded over the last 30 seconds of each exercise. The exercises included running in place, upper arm movements, stepping in place, and obstacle course.

SUMMARY:
This study was designed to evaluate the effectiveness of 12 weeks' home exercise training using the Nintendo ® Wii Fit system in patients with COPD. Following an initial pilot study at one institution to determine the physiological responses to exercise training using the home based interactive computer system, a longitudinal study was performed to evaluate outcomes across several areas. Outcomes were measured at baseline, after 6 weeks of standard care, and after 6 and 12 weeks of home exercise training. Three hospital based pulmonary rehabilitation centers in Connecticut participated in the longitudinal study.

DETAILED DESCRIPTION:
After an initial clinical assessment, which included spirometry or review of recent spirometric data, patients performed an ISWT, as described above. Those who required using supplemental oxygen carried their own tanks. For those who had participated in the pilot study, another ISWT was performed at this time.

Following a 1-hour rest period, baseline outcome assessments were obtained. These included:

1. The Endurance Shuttle Walk Test (ESWT) 9 After an initial warm-up at a slow walk speed, patients walked at an external pace set by an audio source at approximately 85% of their maximal determined by the ISWT. Time at this speed was recorded.
2. Health status. This was measured using the self-reported Chronic Respiratory Questionnaire (CRQ-SR) which has domains of dyspnea, fatigue, emotion and mastery as well as a total score.
3. Dyspnea. This was measured using the 5-point Medical Research Council (MRC) rating.
4. The number of sit-to-stand repetitions in 30 seconds. The patient was seated on a chair without arms and instructed to stand up (without using his/her arms) and then return to the seated position as many times as possible in a 30-second period. This test was first demonstrated by an investigator and then performed by the patient.
5. The number of arm lift repetitions in 60 seconds.11 The subject was instructed to stand and repetitively raise a wooden dowel, from a position resting against the thighs, up to eye level with the arms straight at the elbows, and the return to original position. The maximum number of completed repetitions in 60 s was recorded.

Patients returned after a 6 week non-intervention period when the above-listed outcomes were repeated. They were then given instructions on how to use the Wii Fit unit to perform exercise at home and instructed to perform at least 30 minutes of specified exercises on most days of the week. The required exercises, in sequence, were 1) "Basic Run" (warm up exercise); 2) "Bird's Eye, Bull's-Eye" (mostly upper arm exercise); 3) "Free Step" (mostly lower extremity exercise); 4) "Obstacle Course" (upper and lower extremity exercise); and 5) "Basic Run" (cool down exercise). Additional, ad-lib exercises using this device were allowed. They were instructed to maintain a diary, recording the dates of each session and the total number of minutes devoted to this exercise. Other exercises not based on this system were allowed but not recorded.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent (Approval by the St. Francis Hospital IRB will be required before study initiation)
2. Adults, age > 40 years
3. A clinical diagnosis of COPD, with spirometric confirmation: post-bronchodilator FEV1/FVC < 0.70
4. Moderate, severe and very severe airflow limitation by GOLD criteria.
5. Clinically stable respiratory disease
6. The perceived ability to participate in pulmonary testing and exercise testing
7. COPD, stable state

Exclusion criteria:

1. Women of childbearing potential
2. Asthma
3. Supplemental oxygen use or anticipated oxygen desaturation < 85% at peak exercise (patients who desaturate below 85% on the incremental study will be excluded)
4. Co-morbidity that would interfere with the patient participating in the study, including the exercise testing. Examples include unstable cardiac disease, arthritis, psychological problems that would interfere with participation
5. An exacerbation requiring therapy or any change in maintenance COPD therapy within six weeks of testing
6. A history of a prolonged QT interval
7. Recent exacerbation of COPD

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Oxygen Consumption (VO2) during Wii Exercise | 30 minutes per day

SECONDARY OUTCOMES:
Gender Differences in ESWT performance | 12 weeks
  Measurement comparisons between males and females at baseline, 6 weeks non-intervention, 6 weeks intervention, 12 weeks intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Richard ZuWallack, MD, Principal Investigator — Saint Francis Hospital
Locations (1):
- St Francis Hospital and Medical center, Hartford, Connecticut, United States